CLINICAL TRIAL: NCT00152581
Title: Analysis of the Duration of Combination Therapy That is Necessary for HCV Genotype 1 Eradication
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University College London Hospitals (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01/0277
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2005-12-01 (Estimated); Status verified 2005-09

CONDITIONS: Chronic Hepatitis C, HCV Genotype 1
Keywords: HCV, genotype 1, treatment, HCV kinetics, T-cells
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — peginterferon alfa-2a; Ribavirin

INTERVENTIONS:
Drug: Pegylated interferon-alfa2a (Pegasys); ribavirin

SUMMARY:
Open-label, single centre study evaluating efficacy and viral kinetics of combination PEG-IFNa2a and Ribavirin treatment on CHC genotype 1 patients, administered until viral clearance demonstrated between 4 - 12 weeks, then randomised to further continued combination treatment for one of three defined durations. Followed-up for 24 weeks after treatment cessation.

Objectives:

1. To determine the necessary duration of combination treatment with Pegylated-Interferon alfa2a (PEGASYS) & Ribavirin in Patients infected with genotype 1, in order to achieve viral clearance
2. To identify host factors, which are associated with different patterns of virological response to combination treatment (fast responder, slow responder, non-responder). On this basis, to identify possible predictors for the duration of antiviral treatment.

DETAILED DESCRIPTION:
Forty treatment-naïve patients with chronic hepatitis C, all infected with genotype 1, will be entered into this study. All 40 patients will be started on the same regimen of 180mg Pegylated-Interferon alfa2a (PEGASYS) weekly plus Ribavirin 1000-1200mg daily. HCV RNA in the serum will be monitored by qualitative PCR at treatment weeks 4, 8 and 12. Patients who become HCV RNA negative at any of the above time-points (4,8 or 12), will be randomised into one of three groups to continue the same antiviral regimen for an additional 3 month, 6 month or 9 month period. All these patients will subsequently be followed-up and monitored for a further 6 months after stopping all antiviral treatment.

Treatment will be discontinued for patients who remain persistently HCV RNA positive at treatment week 12 and they will be withdrawn from the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 65
* HCV RNA positive
* HCV genotype 1
* Histologically proven chronic hepatitis
* No previous antiviral treatment

Exclusion Criteria:

* Liver histology showing cirrhosis
* Decompensated liver function
* WCC < 1500/mm3 or platelet count <90,000/mm3
* Co-infection with HIV or HBV/HAV
* Alcohol intake greater than 40 units/week
* Current intravenous drug dependence
* Pregnancy or breast feeding of infants
* Inadequate contraception
* Neuropsychiatric disorder
* Neoplastic disease
* Other significant medical problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2002-04

PRIMARY OUTCOMES:
Sustained virological response (HCV RNA negative) 6 months post-treatment cessation

SECONDARY OUTCOMES:
Hepatic and serum HCV RNA levels as a predictor for treatment duration
HCV-specific T-cell reactivity as a predictor for treatment duration

CONTACTS AND LOCATIONS:
Overall Officials: Nikolai V. Naoumov, MD, Principal Investigator — Institute of Hepatology, University College London
Locations (1):
- Hepatitis Clinic, University College London Hospital, London, United Kingdom